CLINICAL TRIAL: NCT07166289
Title: Parsing Mechanistic Relationships Between Circuits and Negative Valence System Behaviors in Treatment-Resistant Depression With Ultrasound Neuromodulation
Brief Title: Ultrasound Neuromodulation of Circuits and Negative Valence Systems in Treatment-Resistant Depression
Acronym: LIFU CANVAS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2024-011
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Treatment-Resistant Depression
Keywords: Treatment-Resistant Depression; Low-Intensity Focused Ultrasound
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: A sound proof material will be employed to deliver sham stimulation. The operator of the device will be unblinded to the type of intervention (verum vs sham). Participant, assessment team including raters, and staff responsible for evaluation of psychiatric and adverse effects will be blind to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thalamo-Anterior Cingulate Cortex Tract LIFU Sonication (Experimental): An 80-second train of 20-millisecond bursts of ultrasound (0.5 MHz), repeated every 200 milliseconds (400 bursts). It is estimated a 75% tissue attenuation of energy when the ultrasound wave reaches its target, therefore the investigators will set the free-field Intensity Spatial-Peak Pulse-Average (ISPPA) at 9.04 Watt /cm2 or 518 kPascal (to achieve 2.26 Watt/cm2 estimated derated ISPPA). Any modeling of actual energy delivery will be made a posteriori employing BabelBrain® software embedded in the Brainsight® neuronavigation system.
  Interventions: Other: Low-intensity focused ultrasound
- Thalamo- Orbitofrontal Cortex Tract LIFU Sonication (Experimental): An 80-second train of 20-millisecond bursts of ultrasound (0.5 MHz), repeated every 200 milliseconds (400 bursts). It is estimated a 75% tissue attenuation of energy when the ultrasound wave reaches its target, therefore the investigators will set the free-field Intensity Spatial-Peak Pulse-Average (ISPPA) at 9.04 Watt /cm2 or 518 kPascal (to achieve 2.26 Watt/cm2 estimated derated ISPPA). Any modeling of actual energy delivery will be made a posteriori employing BabelBrain® software embedded in the Brainsight® neuronavigation system.
  Interventions: Other: Low-intensity focused ultrasound
- Sham LIFU (Sham Comparator): An 80-second train of 20-millisecond bursts of ultrasound (0.5 MHz), repeated every 200 milliseconds (400 bursts). It is estimated a 75% tissue attenuation of energy when the ultrasound wave reaches its target, therefore the investigators will set the free-field Intensity Spatial-Peak Pulse-Average (ISPPA) at 9.04 Watt /cm2 or 518 kPascal (to achieve 2.26 Watt/cm2 estimated derated ISPPA). Any modeling of actual energy delivery will be made a posteriori employing BabelBrain® software embedded in the Brainsight® neuronavigation system.
  Interventions: Other: Low-intensity focused ultrasound

INTERVENTIONS:
Other: Low-intensity focused ultrasound — 80-second stimulus with an estimated tissue ISSPA=2.26 W/cm2, with (sham) or without (verum) interposition of Sorbothane film

SUMMARY:
Approximately one third of individuals with Major Depressive Disorder (MDD) are considered treatment-resistant, subject to severe disability and risk of suicide, and exhibit symptoms anchored in abnormalities of Research Domain Criteria (RDoC) Negative Valence Systems behavioral processes. In the present study we plan to use low-intensity focused ultrasound in 120 persons with treatment-resistant MDD to modulate deep white matter tracts connecting the thalamus and different regions of the prefrontal cortex reversibly and non-invasively, with the aim of assigning a causal, mechanistic role to large scale brain circuits in the production of those critical behavioral abnormalities. A successful study will help to attain the precise definition of neuromodulation targets for this clinical population in utter need of help.

DETAILED DESCRIPTION:
Approximately one third of individuals with depression are considered treatment-resistant (TRD) and exhibit symptoms anchored in abnormalities of RDoC Negative Valence Systems behavioral processes. For example, anhedonia and rumination contribute to significant impairment in daily functioning, high relapse rates, and a staggering global toll of over 700,000 annual suicides. One reason for inadequate treatment response is our limited understanding of causal mechanisms linking brain circuit function to Negative Valence behavior abnormalities, which impedes the development of precision neuromodulation treatments. The investigators propose to address this problem by using low-intensity focused ultrasound (LIFU), which can noninvasively and reversibly modulate deep brain circuits, to determine the mechanistic relationship between cortico-subcortical circuits and distinct Negative Valence System behaviors including reward processes and rumination. Substantial preliminary evidence suggests that aberrant connectivity between the thalamus and orbitofrontal (OFC) or anterior cingulate (ACC) cortices in the right hemisphere contribute to distinct depression-related RDoC Negative Valence system behavioral changes. In a preliminary clinical trial, which received a non-significant risk determination by the FDA (NCT05697172) the investigators observed safe modulation of deep white matter tracts using LIFU. The investigators now propose to employ advanced structural imaging techniques to tailor modulation targets to each patient's unique anatomy.

The study will involve 120 TRD participants who will receive LIFU and sham stimulation to individually defined white matter tracts connecting thalamus with either OFC (n=60) or ACC (n=60). The investigators will measure resting-state functional magnetic resonance imaging (fMRI) changes, and changes in two behavioral models underlying Negative Valence manifestations (monetary incentive delay and induced rumination tasks). The investigators' hypothesis is that thalamo-OFC and thalamo-ACC hyperconnectivity, historically targeted in neuromodulation techniques useful in TRD, contributes to distortions in distinct behavioral components of the Negative Valence system. This proposal thus has the following Specific Aims: In Aim 1, the investigators will determine the anatomical specificity of LIFU when applied to thalamo-OFC and thalamo-ACC white matter tracts. The investigators predict that LIFU will lead to reduced functional connectivity in the specific cortical regions reached by the modulated white matter bundles. In Aim 2, the investigators will correlate connectivity between thalamus and OFC or ACC, with functional features of distinct behaviors pertaining to the RDoC Negative Valence. Exploratory Aim 3 will establish behavioral correlates of such neural changes. If successful, the present proposal will contribute to understanding clinically meaningful brain-behavior mechanistic relationships by parsing thalamo-prefrontal circuits and RDoC Negative Valence system behaviors. In turn, such definition of targets with a causal role in abnormal behavior processes, could inform precision therapeutic neuromodulation in a psychiatric population in utter need of innovative treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Persons 18-65 years old, with gender and ethnicity recruitment targets including a M:F proportion of 1:2 and White:Black:Hispanic:Native American proportion as close as possible to 8:2:2:1 to reflect the regional epidemiology of TRD (63% White American; 16% African American; 14% Hispanic of any race; 5% Native American),
2. DSM-5-TR diagnosis of MDD as confirmed by MINI structured interview followed by consultation with a board-certified psychiatrist,
3. Evidence of treatment resistance defined as continued MDD symptoms despite any of the following:

   1. two or more adequate (6 week) trials of antidepressants with different mechanisms,
   2. evidence-based psychotherapy,
   3. augmentation agent (lithium, atypical antipsychotic, or T3), or
   4. consideration of ECT or prior ECT nonresponse or intolerance,
4. at least moderate symptoms as indicated by MADRS≥20 upon screening
5. stable treatments including psychotherapy and medication for at least six weeks prior to participation.
6. Fluent English speaker, capable of written consent
7. Consent that random observations of pathology are possible (e.g., brain abnormality seen during imaging)

Exclusion Criteria:

1. Clinical history of at least minor neurocognitive disorder of neurodegenerative origin,
2. PROMIS (Cognitive Function scale) score ≤40 (i.e., mean - 1SD), collected at baseline
3. clinical history of relevant structural pathology of the central nervous system, including Parkinson's disease, multiple sclerosis, and brain malignant neoplasia,
4. uncontrolled diabetes mellitus (as evidenced by a fasting glycemia ≥ 120 mg/dL or hemoglobin A1c ≥ 6.5%) or hypertension (as evidenced by two consecutive readings ≥ 140/90 mmHg) to ensure medical stability, collected at baseline
5. pregnancy or lactation,
6. Has positive test result(s) for alcohol or drugs of abuse (including methadone, opiates, cocaine, amphetamine/methamphetamine, and ecstasy), or substance use disorder including alcohol, stimulants, sedatives, and cannabis exceeding mild severity in the last 6 months,
7. active suicidal ideation (as measured by Suicide-Risk-Assessment-C-SSRS75 "Yes" answers to items 3, 4 or 5 of Suicidal Ideation-Past 1 month section, or any "Yes" answer to any of the items of Suicidal Behavior-Past 3 months section), or any suicide attempt in the last 3 months, collected at baseline
8. MRI contraindications as detected by the MRI Safety Screen, including unwillingness/unable to complete MRI scans
9. medical history indicative of moderate to severe traumatic brain injury as evidenced by history of > 5 minutes of loss of consciousness, or of skull fractures, which in theory could distort LIFU tissue propagation, and
10. a current diagnosis of a psychotic disorder (e.g. schizophrenia, bipolar disorder), an eating disorder (e.g. anorexia or bulimia nervosa), learning disability, or a personality disorder that is considered by the investigator to interfere with the ability of the subject to adhere to the protocol (e.g., narcissistic personality disorder, borderline personality disorder).
11. Has a history of moderate or severe substance or alcohol use disorder according to DSM-5-TR
12. Use of benzodiazepines or anticonvulsants in the 7 days prior to screening
13. Medical, psychiatric, or other conditions that restrict the patient's following abilities: to interpret the study information, to give informed consent, to adhere to the rules of the protocol, or to complete the study.
14. No reliable method of communication (i.e., no access to internet or phone connection)
15. Prescription of a medication outside of the accepted range, as determined by best clinical practices and current research
16. Unwillingness or inability to complete any of the major aspects of the study protocol
17. Non-correctable vision or hearing problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2030-04 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Post-Sonication Changes in Functional Connectivity | Pre- vs up to 30 minutes post-sonication or sham intervention.
  Changes in resting-state functional (fMRI) connectivity (FC) between thalamus and either Anterior Cingulate (ACC) or Orbitofrontal (OFC) cortices after LIFU or Sham stimulation.
Post-Sonication Changes in Reward and Repetitive Mentation | Up to 30 minutes post-sonication vs sham intervention
  Changes in BOLD activation of either Anterior Cingulate (ACC) or Orbitofrontal Cortex (OFC) during Monetary Incentive Delay and Induced Rumination Tasks corresponding to changes in reward and repetitive thinking, respectively.

SECONDARY OUTCOMES:
Post-Sonication Changes in Functional Connectivity and Anhedonic and Ruminative Symptoms | Pre- vs up to 30 minutes post-sonication
  Changes in functional connectivity of thalamo-frontal and thalamo-anteiror cingulate regions and the correlation to changes in Snaith-Hamilton Pleasure Scale scores (minimum score: 0; maximum score: 14; lower scores mean better outcomes) and Brief State Rumination Inventory Scores (minimum value: 0; maximum value: 25; lower scores mean better outcomes) to evaluate anhedonic and ruminative symptoms respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No